CLINICAL TRIAL: NCT05479851
Title: ORCA: Opportunities to Raise Cancer Awareness After Referral: Survey of Patient Views
Acronym: ORCA
Status: Completed | Type: Observational
Sponsor: King's College London (Other)
Collaborators: Guy's and St Thomas' NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 303199
Record Dates: First submitted 2022-04-19; First posted 2022-07-29 (Actual); Last update posted 2023-06-15 (Actual); Status verified 2023-06

CONDITIONS: Cancer
Keywords: Cancer early diagnosis; Cancer awareness; Cancer risk reduction behaviour; Health Behaviour
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- UK National Health Service Patient Postal Survey Participants: Patients who have agreed to participate in the study after receiving a postal invitation

SUMMARY:
The purpose of this study is to investigate what patients think about increasing provision of advice about how to detect cancer early and how to reduce their future cancer risk after they are discharged from a two-week wait referral pathway for suspected cancer. This study will send a postal survey to patients living in the UK who were recently referred onto the suspected cancer pathway and were discharged without a cancer diagnosis (i.e. a negative diagnosis). Patients will be presented with different types of support and patients' views of the burden, benefits, understanding and perceived effectiveness of each one will be measured.

DETAILED DESCRIPTION:
In England, over 2 million patients are referred each year on urgent two-week wait (TWW) pathways to rule-out cancer of a single anatomical site. Referrals have increased by around 10% per year since 2015 (with the exception of 2020, due to the COVID-19 pandemic). The vast majority of those referred (93%) do not have cancer diagnosed. There is mounting evidence that patients who have previously experienced a symptom that after investigation turned out to be benign, often delay seeking help for subsequent symptoms. This is thought to occur because of over-reassurance from the previous 'all-clear' result leading to subsequent symptoms being interpreted as benign (extending the appraisal interval), concern about appearing hypochondriacal, not wanting to further bother the doctor or about the appropriate next actions. This is likely to be compounded by the impact of COVID-19 on help-seeking decisions and has implications for service provision. There may be scope to provide tailored support to those who are initially discharged without a cancer diagnosis to avoid missing cancers at other anatomical sites and to ensure subsequent cancers are diagnosed in a timely manner, at an early stage, or even prevented. For instance, patients could be offered information on common cancer signs, when/how to seek help for ongoing or new symptoms, facilitation to take part in cancer screening, and preventative advice. Indeed, referral for suspected cancer may be an under-utilised 'teachable moment' when people are more responsive and receptive to health information. There is currently a lack of support for those with a negative diagnosis after a TWW referral. Qualitative work indicates that there is currently no standardised approach to the information patients receive from healthcare professionals about future cancer risk or how to respond to new or recurring symptoms. It is important to assess feasibility and acceptability of interventions prior to evaluation of effectiveness. This allows implementation strategies to be incorporated into the design of interventions that will increase adoption and sustainment as well as being appropriate to the setting, providers and recipients. Yet at present it is not known what the feasibility and acceptability is of interventions linked to the TWW pathway. The objective of the proposed research is to obtain this information.

ELIGIBILITY:
Inclusion Criteria:

1. Adults >18 years old
2. Referred through the two-week wait pathway for suspected cancer
3. Received a negative diagnosis (i.e. informed of a 'ruling out of cancer' according to the new 28-day faster diagnosis standard) within the past 1-3 months

Exclusion Criteria:

1. Adults who have been diagnosed with cancer
2. Adults who have not yet been informed of their results from their urgent referral

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adults >18 years old who have been referred through the two-week wait pathway for suspected cancer, and who have received a negative diagnosis (i.e. informed of a 'ruling out of cancer' according to the new 28-day faster diagnosis standard).
Sampling Method: Non-Probability Sample
Enrollment: 406 (Actual)
Dates: Start 2022-10-07 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2023-03-31 (Actual)

PRIMARY OUTCOMES:
Participants' prospective acceptability ratings of different types of cancer advice and support interventions using a thirteen-item scale | cross sectional questionnaire to be completed 1-3 months after urgent referral
  Prospective acceptability (perceived acceptability prior to intervention participation) of different cancer advice and support interventions, will be compared using scores obtained from a 13-item scale reflecting the domains of the Theoretical Framework of Acceptability (Scott et al 2021).

SECONDARY OUTCOMES:
Proportions of participants willing to receive each type of advice/ support, after discharge from a two week wait (urgent referral) pathway | cross sectional questionnaire to be completed 1-3 months after urgent referral
  Comparison of the willingness of participants from different two week wait pathways to receive different types of advice/ support. Willingness will be assessed using a one-item measure (Stevens et al 2019, Prev Med; Stevens et al, 2019, Lung Cancer).

CONTACTS AND LOCATIONS:
Locations (1):
- King's College London, London, Surrey, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
We will obtain consent for electronic copies of anonymised non-personally identifiable data (e.g. questionnaire responses) to be archived, shared and available for secondary analysis via a data sharing repository (e.g. King's College London (KCL) data repository). Data will be uploaded to the repository upon acceptance of publication or within 3 months of the end of the funding, whichever occurs earliest.
Time Frame: Data will be uploaded to the repository upon acceptance of publication or within 3 months of the end of the funding, whichever occurs earliest.
Access Criteria: Anonymous questionnaire data will be available for use via the repository by other researchers if they have further ethical approval to re-use the data.

REFERENCES:
- [Background] Scott SE, Rauf B, Waller J. "Whilst you are here..." Acceptability of providing advice about screening and early detection of other cancers as part of the breast cancer screening programme. Health Expect. 2021 Oct;24(5):1868-1878. doi: 10.1111/hex.13330. Epub 2021 Aug 8. PMID 34369071
- [Background] Stevens C, Vrinten C, Smith SG, Waller J, Beeken RJ. Acceptability of receiving lifestyle advice at cervical, breast and bowel cancer screening. Prev Med. 2019 Mar;120:19-25. doi: 10.1016/j.ypmed.2018.12.005. Epub 2018 Dec 19. PMID 30578909
- [Background] Stevens C, Smith SG, Quaife SL, Vrinten C, Waller J, Beeken RJ. Interest in lifestyle advice at lung cancer screening: Determinants and preferences. Lung Cancer. 2019 Feb;128:1-5. doi: 10.1016/j.lungcan.2018.11.036. Epub 2018 Nov 27. PMID 30642439